CLINICAL TRIAL: NCT06734312
Title: Gastric Fundal Mucosal Ablation for Weight Management in Patients Stopping Glucagon-like Peptide-1 Receptor Agonists
Brief Title: MAINTAIN (Mucosal AblatIoN Therapy After INcretins)
Acronym: MAINTAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Christopher McGowan (Other)
Responsible Party: Sponsor-Investigator, Dr. Christopher McGowan, Co-Founder/Co-CEO/Chief Medical Officer, True You Weight Loss
Organization: True You Weight Loss (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-004
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions; Obesity and Overweight; Obesity Prevention; Obesity Recidivism; GLP-1; Ablation Techniques
Keywords: obesity; obesity and overweight; endoscopic bariatric therapy; ablation; gastric mucosal ablation; GMA; GFMA; glp-1; weight loss medications; weight loss; semaglutide; tirzepatide; hunger; appetite
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gastric Fundal Mucosal Ablation (GFMA) following discontinuation of GLP-1 therapy (Experimental): Subjects will undergo endoscopic Gastric Fundal Mucosal Ablation (GFMA) following following discontinuation of GLP-1 therapy. This will be performed by an experienced endoscopist specialized in bariatric endoscopy in a single endoscopic session.
  Interventions: Device: Gastric Fundal Mucosal Ablation (GFMA)

INTERVENTIONS:
Device: Gastric Fundal Mucosal Ablation (GFMA) — Endoscopic Gastric Fundal Mucosal Ablation (GFMA) after discontinuation of GLP-1 therapy

SUMMARY:
The purpose of this study is to assess the effect of gastric fundal mucosal ablation (GFMA) on weight trajectory following discontinuation of once-weekly semaglutide or tirzepatide in adults with obesity. In this study, GFMA will be performed on patients who have experienced > 10% weight loss with GLP-1 therapy and who plan to discontinue use of GLP-1 medications for the duration of the study.

DETAILED DESCRIPTION:
Obesity is a multifactorial, chronic, and progressive disease of pandemic proportions. Incretin mimetics , such as semaglutide and tirzepatide, induce weight loss in adults with obesity, while also improving weight-related medical conditions, such as cardiac and renal disease. The beneficial effects on weight and metabolism require the continued presence of these medications, which have a half-life of approximately five to seven days. This concept was substantially illustrated in the STEP4 and SURMOUNT4 randomized controlled trials. In the STEP4 trial, adults with obesity were treated with semaglutide for a 20-week run-in, losing 10.6% of body weight, thereafter randomized 2:1 to continued semaglutide use vs placebo. Over the subsequent 48 weeks, the semaglutide arm lost an additional 7.9% of original body weight, whereas the placebo arm saw two-thirds the lost weight return. In the SURMOUNT-4 trial, adults with obesity were treated with tirzepatide for a 36-week run-in period, losing 20.9% of body weight, thereafter, randomized 1:1 for continued treatment or placebo. Over the subsequent 52 weeks, the treatment arm lost an additional 5.5% of body weight, whereas the placebo arm saw a return of approximately half the weight that had been lost. These observations present challenges for long-term obesity management when confronted by multiple reports showing high rates of discontinuation of incretin mimetics soon after initiation. These observations present challenges for long-term obesity management when confronted by multiple reports showing high rates of discontinuation of incretin mimetics soon after initiation. Gastric fundal mucosal ablation (GFMA) is a novel endoscopic approach to control appetite which uses hybrid argon plasma coagulation (HybridAPC) to ablate the superficial tissue of the gastric fundus to induce cell death and fibrotic remodeling. In an early safety and feasibility study of ten adults with obesity, GFMA reduced circulating levels of the only known hunger hormone in humans, ghrelin. This led to a measured suppression of inter-meal hunger and cravings, as well as improved confidence in the ability to resist cravings. In addition to reducing ghrelin-producing cell population within the fundus, GFMA induced significant fundal fibrin deposition. This resulted in a stiffer, less compliant fundus, reducing maximum tolerated volume of a standardized nutrient drink test, enhancing intra-meal satiation. Given that GFMA induces appetite control through both visceroceptive and hormonal mechanism, much like incretin mimetics, we hypothesize that GFMA can prevent or limit weight recurrence in adults who have stopped these medications after successful obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 21-65
2. Body mass Index (BMI) ≥30 kilograms per square meter (kg/m²), or ≤45 kg/m²
3. Observed ≥ 10% TBWL with semaglutide or tirzepatide use for primary obesity therapy
4. Subject did not experience >50% weight recurrence since discontinuation of semaglutide or tirzepatide
5. Maintained a stable dose of semaglutide or tirzepatide for a minimum of 12 weeks
6. Have recently discontinued or are planning to discontinue semaglutide or tirzepatide (≤ 24 weeks from last dose to time of study procedure)
7. No previous medical history of diabetes mellitus
8. Willing and able to participate in the study procedures
9. Understand and voluntarily sign the informed consent

Exclusion Criteria:

1. Known diagnosis of type I or type II diabetes or a Hemoglobin A1c > 6.5% at time of screening
2. Use of GLP-1 or GLP-1/GIP medication for the treatment of diabetes, rather than obesity.
3. Use of anticoagulation, antithrombotic agents, and/or NSAIDs that cannot be discontinued for a minimum of 12 weeks
4. Known bleeding diathesis that cannot be corrected through medical means.
5. History of decompensated end-organ disease
6. Unwillingness to abstain from the use of incretin mimetics during the study duration.
7. Unwillingness to abstain from the use of tobacco during the study duration
8. Patients on any medications or supplements including those that may influence cholecystokinin (CCK), glucose, growth hormone, insulin and/or somatostatin levels
9. History of any stomach manipulation (including repair of hiatal hernia or fundoplication) deemed unsafe by PI for GFMA
10. Active disordered eating
11. Patients who do not give their consent to the enrollment in the study or are incompetent, unconscious or unable to express their consent for any reason
12. Known diagnosis of gastroparesis or functional dyspepsia
13. Patients who are pregnant, who plan to become pregnant during study duration, or patients of child-bearing potential who refuse effective birth control methods (as approved by PI)
14. Active H. pylori infection or history of H pylori without treatment and confirmation of eradication
15. Active gastric ulceration.
16. Use of concomitant medications known to induce weight loss (including but not limited to liraglutide, phentermine, phentermine/topiramate, bupropion/naltrexone, metformin)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Total Body Weight Loss (TBWL) from Baseline | 12 months
  Measure percent change in total body weight over time following endoscopic GFMA. TBWL = pre-op weight - post op body weight. % TBWL is the fraction of body weight expressed in percentage term

SECONDARY OUTCOMES:
Rate of Adverse Events (AE) | Month 1, Month 2, Month 3, Month 4, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Occurrence of Adverse Events along with AE Type, severity, and relationship to treatment.
Quality of Life Assessment | 1 Month, 2 Months, 3 Months, 6 Months, 12 Months
  Baseline quality of life assessment scores compared to follow-up quality of life assessment scores. Quality of life score assessed and measured by the Impact of Weight on Quality of Life-Lite questionnaire. Scoring for the questionnaire ranges from 0 (minimum) to 100 (maximum). Higher scores for the Impact of Weight on Quality of Life-lite questionnaire indicates higher quality of life.
Quality of Life Assessment | 1 Month, 2 Months, 3 Months, 6 Months, 12 Months
  Baseline quality of life assessment scores compared to follow-up quality of life assessment scores. Quality of life score assessed and measured by the 36-Item Short Form Survey. Scoring for the questionnaire ranges from 0 (minimum) to 100 (maximum). Higher scores on the 36-Item Short Form Survey questionnaire indicates higher quality of life.
Appetite and Hunger Assessment | Month 1, Month 2, Month 3, Month 6, Month 12
  Baseline appetite and hunger assessment scores compared to follow-up appetite and hunger assessment scores. Appetite and hunger assessed and measured by the DAILY EATS questionnaire, which contains a numerical rating scale of 0-10 for each its 5 items. A higher score indicates greater hunger and appetite. A reduction in DAILY EATS score from baseline indicates a decrease in hunger and appetite levels, which is considered a positive outcome.
Percent Change in Total Body Weight Loss (TBWL) from Baseline | Month 1, Month 3, Month 6, Month 9
  Measure percent change in total body weight over time following endoscopic GFMA. TBWL = pre-op weight - post op body weight. % TBWL is the fraction of body weight expressed in percentage term
Change in Body Mass Index (BMI) from Baseline | Month 1, Month 3, Month 6, Month 9, Month 12
  Measure change in body mass index over time following endoscopic GFMA. BMI=(Weight in kg)/((Height in meters) ^2)
Percent Weight Recurrence from Baseline | Month 1, Month 3, Month 6, Month 9, Month 12
  Measure percent recurrence in weight following endoscopic GFMA following discontinuation of semaglutide or tirzepatide.
  % Weight recurrence = % of weight lost from semaglutide or tirzepatide that recurs after discontinuation
Measured Proportion of Patients with weight recurrence | 6 Months, 12 Months
  Measure percentage of patients with weight recurrence between <0%, 0-19.9%, 20-39.9%, 40-59.9%, 60-79.9%, 80-99.9%, vs 100% or more after GFMA.
Eating Behavior and Weight Management Self-Efficacy Assessment | Month 1, Month 2, Month 3, Month 6, Month 12
  Baseline eating behavior and weight management self-efficacy assessment scores compared to follow-up eating behavior and weight management self-efficacy scores measured by the WEL-SF questionnaire. WEL-SF is scored on a scale of 0-80 and includes 8 items measuring eating self-efficacy, which is the confidence one has in their ability to resist overeating. Higher WEL-SF scores indicate greater eating behavior self-efficacy and control. An increase in WEL-SF scores from baseline reflects an improvement in eating self-efficacy and is considered a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McGowan, MD, MSCR, Principal Investigator — True You Weight Loss
Locations (1):
- True You Weight Loss, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumbhari V, Lehmann S, Schlichting N, Heinrich M, Kullnick Y, Retschlag U, Enderle M, Dietrich A, Khashab MA, Kalloo AN, Oberbach A. Gastric mucosal devitalization is safe and effective in reducing body weight and visceral adiposity in a porcine model. Gastrointest Endosc. 2018 Jul;88(1):175-184.e1. doi: 10.1016/j.gie.2018.02.022. Epub 2018 Feb 22. PMID 29476845
- [Background] Wilding JPH, Batterham RL, Davies M, Van Gaal LF, Kandler K, Konakli K, Lingvay I, McGowan BM, Oral TK, Rosenstock J, Wadden TA, Wharton S, Yokote K, Kushner RF; STEP 1 Study Group. Weight regain and cardiometabolic effects after withdrawal of semaglutide: The STEP 1 trial extension. Diabetes Obes Metab. 2022 Aug;24(8):1553-1564. doi: 10.1111/dom.14725. Epub 2022 May 19. PMID 35441470
- [Background] Popoviciu MS, Paduraru L, Yahya G, Metwally K, Cavalu S. Emerging Role of GLP-1 Agonists in Obesity: A Comprehensive Review of Randomised Controlled Trials. Int J Mol Sci. 2023 Jun 21;24(13):10449. doi: 10.3390/ijms241310449. PMID 37445623